CLINICAL TRIAL: NCT04157673
Title: Imagine to Remember: Improving Medication Adherence in Pre- and Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Leonard Epstein, SUNY Distinguished Professor and Division Chief, Behavioral Medicine, State University of New York at Buffalo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FWA00008824
Record Dates: First submitted 2019-11-06; First posted 2019-11-08 (Actual); Results first posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Medication Adherence
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Intervention Model Description: This study is a multiple-baseline single subject design; participants will be randomized to intervention at 6-week, 8-week, or 10-week.
Masking Description: Participants will not be informed of the group that they are randomly assigned until the completion of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Episodic Future Thinking introduced at 6 weeks (Experimental): The intervention being researched is called episodic future thinking (EFT), which consists of imagining specific instances of one's future. In this study, participants will engage in EFT focused on imagining taking one's medication, guided by a research staff member in their intervention sessions in addition to weekly check-in calls across an 8-week period following a 6-week, 8-week or 10-week baseline period. The research staff member will conduct the intervention session using a semi-structured interview format in which they work to identify situations in which the participant encounters challenges with taking their medication and will ask questions to prompt the participant to imagine what successful medication adherence would consist of. Sessions may also involve imagining positive events resulting from successful medication adherence and the details surrounding those events.
  Interventions: Behavioral: Episodic Future Thinking

INTERVENTIONS:
Behavioral: Episodic Future Thinking — This intervention involves participants engaging in episodic future thinking in order to improve their medication adherence and overall prospective thinking ability. This intervention will be introduced following a 6-week, 8-week or 10-week baseline period.

SUMMARY:
Determine if an intervention consisting of future-thinking improves different facets of memory/executive function and/or decision-making.

DETAILED DESCRIPTION:
The aim of this study is to determine if a cognitive intervention is an efficacious method for improving medication adherence in adults with prediabetes or type 2 diabetes. Participants in this study will complete assessment sessions, as well as intervention sessions over a 15 week period. During this time, medication adherence will be monitored using a MEMS cap. The investigators hypothesize that, following the cognitive intervention, there will be improvements in participants' medication adherence, as well as in facets of memory.

ELIGIBILITY:
Inclusion Criteria:

Adults over the age of 18 with prediabetes or Type 2 Diabetes currently prescribed at least one oral medication for blood glucose regulation, or for related comorbidities e.g., hypertension, hyperlipidemia, and are relatively non-adherent to taking them (< 80% of prescribed doses taken), but are motivated and/or have the intent to better comply with their medication regimen, will be studied.

Prediabetes and Type 2 Diabetes: Participants must have a diagnosis of prediabetes or Type 2 Diabetes within the last 2 years or meet criteria for prediabetes or Type 2 Diabetes. The American Diabetes Association guidelines (Group, 2003) defines prediabetes and Type 2 Diabetes as Fasting Plasma Glucose (FPG) 100mg/dl or greater, 2h glucose 140mg/dl or greater after Oral Glucose Tolerance Test (OGTT), or hemoglobin A1c (HbA1c) of approximately 5.4% or greater.

Exclusion Criteria:

Pregnancy: Women who are pregnant or lactating will be excluded from participation.

Substance use, abuse, or dependence: Individuals that currently have problems with substance dependence, addiction, or problematic substance use that would limit participation (e.g., binge drinkers, alcoholics, daily stimulant/opiate users) will be excluded.

Conditions that affect adherence: Participants should not have a condition that would limit participation which include medical conditions that would affect individuals' ability to use the computer for prolonged period of time; leave the individual unable to ambulate; unmanaged psychiatric disorder (e.g., depression, anxiety, attention deficit hyperactivity disorder, schizophrenia), cognitive impairment that would impact memory (e.g., symptomatic concussion), or an intellectual impairment that would impact study adherence. Additionally, participants should be able to attend to all intervention sessions. If a participant is not able to make most sessions (e.g. participant is out of town during most of the study for work or vacation travel), they may be excluded from the study Prior participation in similar studies: Individuals who have recently participated in a laboratory study using similar methods may also be excluded.

Use of medication adherence aids: individuals who currently use aids to assist with medication adherence (e.g., pill organizers, reminder apps)may be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University at Buffalo, Department of Pediatrics, Division of Behavioral Medicine, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants completed a screening session prior to baseline period (n =7), in which they completed baseline measures of delay discounting, prospective memory tasks, and medication adherence. 4 participants were eligible and were assigned a baseline time-length (6-, 8- or 10- weeks). Participants were randomized to a baseline time length prior to baseline measurement. Data will be reported in aggregate, rather than by arm (baseline length) due to confidentiality concerns (as n = 1 for 2 arms).
Groups:
- Episodic Future Thinking: The intervention being researched is called episodic future thinking (EFT), which consists of imagining specific instances of one's future. In this study, participants will engage in EFT focused on imagining taking one's medication, guided by a research staff member in their intervention sessions in addition to weekly check-in calls across an 8-week period following a 6-week, 8-week or 10-week baseline period. The research staff member will conduct the intervention session using a semi-structured interview format in which they work to identify situations in which the participant encounters challenges with taking their medication and will ask questions to prompt the participant to imagine what successful medication adherence would consist of. Sessions may also involve imagining positive events resulting from successful medication adherence and the details surrounding those events.
  Episodic Future Thinking: This intervention involves participants engaging in episodic future thinking in order to improve their medication adherence and overall prospective thinking ability. This intervention will be introduced following a 6-week, 8-week or 10-week baseline period.
Period: Overall Study
Arm/Group | Episodic Future Thinking
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Episodic Future Thinking: The intervention being researched is called episodic future thinking (EFT), which consists of imagining specific instances of one's future. In this study, participants will engage in EFT focused on imagining taking one's medication, guided by a research staff member in their intervention sessions in addition to weekly check-in calls across an 8-week period following a 6-week, 8-week or 10-week baseline period. The research staff member will conduct the intervention session using a semi-structured interview format in which they work to identify situations in which the participant encounters challenges with taking their medication and will ask questions to prompt the participant to imagine what successful medication adherence would consist of. Sessions may also involve imagining positive events resulting from successful medication adherence and the details surrounding those events.
  Episodic Future Thinking: This intervention involves participants engaging in episodic future thinking in order to improve their medication adherence and overall prospective thinking ability. This intervention will be introduced following a 6-week, 8-week or 10-week baseline period.
  Data will be reported in aggregate, rather than by arm (baseline length) due to confidentiality concerns (as n = 1 for 2 arms).
Arm/Group | Episodic Future Thinking
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 1
  Female | 2
  Non-binary | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4
Baseline Medication Adherence [Mean (Full Range); unit: Percent] — Baseline Medication adherence, measured over the first week for all participants.
  Percent | 57.1 [7.1 to 92.9]

OUTCOME MEASURES:

1. Primary Outcome: Medication Adherence
Description: The investigators will measure medication adherence using a medication event monitoring system (MEMS) that measured the frequency and time the medication bottle is opened. Percent adherence was calculated [(Quantity of pills dispensed - remaining)/(quantity prescribed per day*days since last refill)] *100. Percent change was calculated from the last week of baseline to the first week of EFT and the last week of EFT
Time Frame: 15 weeks
Population: Data will be reported in aggregate, rather than by arm (baseline length) due to confidentiality concerns (as n = 1 for 2 arms).
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Episodic Future Thinking
Number analyzed (Participants) | 4
percent change
  Last week of Baseline to first week of treatment | 34 (28)
  Last week of baseline to last week of treatment | 42 (36)
Statistical Analysis 1: Comparison: Episodic Future Thinking; Statistical analysis to support visual inspection of the multiple-baseline graphs included the phase changes from baseline to Episodic future thinking treatment. Phase changes were assessed using mixed model with fixed effects of level and trend for baseline phase and random effects for level and trend for treatment phase; Test type: Superiority; p = 0.0002, Mixed Models Analysis — This is the overall treatment effect from the mixed model. p-value threshold set at p = 0.05

2. Primary Outcome: Prospective Memory
Description: Prospective memory ability will be assessed using an event-based version of the virtual week task. This is a computer-based task in which participants are asked to completed different events at specified times in the style of a board game. For the event-based task, participants were asked to complete an extra mouse click when certain words appeared on the screen. Possible scores ranged from 0 - 8 with higher scores being indicative of better prospective memory.
Time Frame: 15 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number correct
Arm/Group | Episodic Future Thinking
Number analyzed (Participants) | 4
Number correct | 0.083 (0.104)
Statistical Analysis 1: Comparison: Episodic Future Thinking; [analysis description as in outcome 1, analysis 1]; Test type: Other — Effect size of mean differences; Mean Difference (Final Values) = 2.75, Standard Deviation 3.78 — Cohen's d effect size = 0.73

3. Secondary Outcome: Delay Discounting
Description: Delay Discounting will be assessed using an adjusting amount task where choices will be present between a larger, delayed amount of money ($100) and a smaller, immediate amount. The smaller, immediate amount will begin at $50 on the first trial and will be adjusted following each trial. Participants cues created during treatment will be displayed during the task. To calculate discount rates area under the curve will be used, in which normalized values of delayed reward and normalized values of delay are used, resulting in values from 0.0 (all immediate choices) and 1.0 (all delayed choices) result. Units are proportion of maximum delayed reward x proportion of maximum delay.
Time Frame: 15 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: proportion max reward x proportion delay
Arm/Group | Episodic Future Thinking
Number analyzed (Participants) | 4
proportion max reward x proportion delay | 0.355 (0.295)
Statistical Analysis 1: Comparison: Episodic Future Thinking; Test type: Other — Effect size of mean pre-post differences; Mean Difference (Final Values) = 0.355, Standard Deviation 0.295 — cohen's d effect size for mean differences pre to post-treatment = 1.20

ADVERSE EVENTS:
Time Frame: 15 weeks
Arm/Group | Episodic Future Thinking
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-22): https://cdn.clinicaltrials.gov/large-docs/73/NCT04157673/Prot_SAP_000.pdf
  • Informed Consent Form (2020-07-22): https://cdn.clinicaltrials.gov/large-docs/73/NCT04157673/ICF_001.pdf